## Randomized, Controlled Cross-over Comparison of Cannabidiol to Oral Opioid for Postoperative Photorefractive Keratectomy Pain Control

## 2. Statistical Analysis Plan

JASP 0.19.0 will be used to calculate baseline statistics and cohort demographics such as age, sex, and initial vision. Fisher test will be used to ensure equal allocation between groups and drug treatments. Multiple Repeated Measures ANOVA will be used to test for differences between vision, pain, and other secondary outcomes after using each drug. For survey outcomes, no comparison was made between drugs because outcomes were binocular and associated with use of both drugs. Alpha will be 0.05 for this study. Beta was estimated approximately 0.80 based on a sample size of 70 units (35 patients each eye).